CLINICAL TRIAL: NCT03317860
Title: Improving Measurement and Treatment of Post-stroke Neglect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: N2420-W; 1IK2RX002420-01A2 (NIH)
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: perceptual disorders; cerebrovascular disorders; neurobehavioral manifestations; neurologic manifestations; neglect; non-invasive brain stimulation; rehabilitation; tDCS; paresis
MeSH Terms: conditions — Stroke; Perceptual Disorders; Cerebrovascular Disorders; Neurobehavioral Manifestations; Neurologic Manifestations; Paresis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will receive both conditions (active and sham transcranial direct current stimulation paired with arm rehabilitation training [repetitive task-specific practice]) in this cross-over design study. Individuals will be randomized to determine which condition they receive first and the participant and treatment therapist and assessor will be blinded to the order that the interventions are delivered. The PI will oversee randomization so that each patient is randomized and assigned a unique five digit code. When this code is entered on the tDCS device, the device will automatically assign the patient to receive either real or sham stimulation. Because the sham stimulation provides a ramp up/ramp down stimulation for 15 seconds at the start and end of the session the participant may perceive the sham stimulation as active stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham tDCS plus RTP (Sham Comparator): Single session of bilateral sham parietal cortex tDCS (for 30 minutes) paired with repetitive task-specific practice (RTP)
  Interventions: Device: Sham tDCS
- Active tDCS plus RTP (Active Comparator): Single session of bilateral active parietal cortex tDCS (2.0 mA for 30 minutes) paired with repetitive task-specific practice (RTP)
  Interventions: Device: Active tDCS

INTERVENTIONS:
Device: Sham tDCS — Sham tDCS will be delivered for 30 minutes in conjunction with repetitive task-specific practice for the arm/hand. tDCS is a form of noninvasive brain stimulation. Electrodes will be placed on the scalp but in the sham condition they will not deliver direct current (2mA). Sham tDCS will be delivered for 30 minutes in conjunction with repetitive task-specific practice for the arm/hand.
  Repetitive task-specific practice (RTP). Participants will practice using their paretic arm/hand to complete functional movements during the 30 minute train
  Other Names: noninvasive brain stimulation, transcranial direct current stimulation
  Arms: Sham tDCS plus RTP
Device: Active tDCS — Sham tDCS will be delivered for 30 minutes in conjunction with repetitive task-specific practice for the arm/hand. tDCS is a form of noninvasive brain stimulation. Electrodes will be placed on the scalp but in the sham condition they will not deliver direct current (2mA). Sham tDCS will be delivered for 30 minutes in conjunction with repetitive task-specific practice for the arm/hand.
  Repetitive task-specific practice (RTP). Participants will practice using their paretic arm/hand to complete functional movements during the 30 minute train
  Other Names: noninvasive brain stimulation, transcranial direct current stimulation
  Arms: Active tDCS plus RTP

SUMMARY:
This study examines how to best assess and treat post-stroke neglect. This study will examine the preliminary effects of an innovative intervention (repetitive task-specific practice + transcranial direct current stimulation) for individuals with neglect. This study will also determine whether items from various neglect assessments can be combined to establish a more comprehensive neglect measure.

DETAILED DESCRIPTION:
It is very common for stroke survivors to have difficulty attending to one side of their body or space (neglect). Stroke survivors with neglect not only demonstrate impairments in attention but they also experience motor impairment. These individuals also have an imbalance in excitation in the brain. This study will examine the preliminary effects of non-invasive brain stimulation (transcranial direct current stimulation, tDCS) combined with arm rehabilitation training (repetitive task-specific practice, RTP) for individuals with neglect following stroke. The investigators will examine the effects of the intervention on brain excitability, upper extremity motor impairment, and attentional impairment. This study will also examine assessment of neglect. There are many clinical assessments designed to assess neglect; however, it is unknown whether items from some of the most commonly used assessments are able to effectively measure neglect or whether items from these assessments can be combined. Clinicians rely on clinical assessments to inform treatment and document patient progress. Therefore, it is important that investigators more closely examine these existing assessments.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke 3 months post stroke.
* Fugl-Meyer Upper Extremity (FMA-Upper Extremity) score between 20-56/60
* Inducible motor evoked potential (MEP) of the abductor pollicis brevis (APB) on the paretic stimulation (TMS)
* Demonstrate the presence of unilateral neglect (Virtual Reality Lateralized Attention Test score <18)

Exclusion Criteria:

* History of cortical hemorrhagic stroke
* Presence of any MRI, TMS, tDCS risk factors including:

  * history of seizures
  * history of brain tumor
  * hardware in skull or spine (e.g. coils, clips)
  * implantable medical device (e.g. pacemaker)
  * metal in body (not compatible with MRI)
  * pregnancy
* Severe spasticity (Modified Ashworth Scale score 3)
* Severe aphasia or cognitive impairment limiting participants' comprehension (National Institutes of Health Stroke Scale Level of Consciousness Commands Item score 1 or Best Language Item score 2)
* Unable to travel to UE Motor Function Laboratory at the Center for Rehabilitation Research in Neurological Conditions (a collaborative, MOU approved, research center Ralph H. Johnson VA Medical Center and the Medical University of South Carolina) for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2018-07-02 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in excitability of fronto-parietal connectivity | Participants will be assessed at baseline and 30 minutes later
  Excitability of fronto-parietal connectivity measured by paired pulse twin coil transcranial magnetic stimulation (TMS) test. In each session, the difference in excitability of fronto-parietal connectivity between pre and post stimulation will be measured.

SECONDARY OUTCOMES:
Change in upper extremity kinematics | Participants will be assessed at baseline and 30 minutes later
  A kinematic assessment will be conducted to assess changes in motor impairment.
Change on Behavioral Inattention Test | Participants will be assessed at baseline and 1.5 hours later (immediately following experimental condition)
  A neglect assessment (conventional subtests) will be conducted to assess changes in attentional impairment. Total scores range from 0-146 with lower scores indicating greater impairment.

OTHER OUTCOMES:
Catherine Bergego Scale | Participants in the cross-sectional study will be assessed at baseline.
  This neglect assessment will be administered to examine the impact of neglect on performance of daily activities. Total scores range from 0-30 with higher scores indicating greater impairment.
Behavioral Inattention Test | Participants in the cross-sectional study will be assessed at baseline.
  This neglect assessment (behavioral subtests) will be administered to examine the impact of neglect on performance of daily activities. Total scores range from 0-81 with lower scores indicating greater impairment.
Naturalistic Action Test | Participants in the cross-sectional study will be assessed at baseline.
  This neglect assessment will be administered to examine the impact of neglect on performance of daily activities. Each item has a score of 0-6 with lower scores indicating greater impairment. The Lateralized Attention Score (LAS) is difference between the contralateral and ipsilateral proportion of items. Higher LAS scores indicate greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Emily S. Grattan, PhD MS BS, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Longley V, Hazelton C, Heal C, Pollock A, Woodward-Nutt K, Mitchell C, Pobric G, Vail A, Bowen A. Non-pharmacological interventions for spatial neglect or inattention following stroke and other non-progressive brain injury. Cochrane Database Syst Rev. 2021 Jul 1;7(7):CD003586. doi: 10.1002/14651858.CD003586.pub4. PMID 34196963